CLINICAL TRIAL: NCT00764634
Title: A Phase 2, Randomized, Double Blind, Placebo-Controlled, Multicenter Study to Evaluate Safety, Dosing Schedule and Antibody Kinetics of Recombinant Botulinum Vaccine A/B, rBV A/B-40, in Healthy Adults
Brief Title: Double Blind, Safety and Immunogenicity Study of Recombinant Botulinum Vaccine A/B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: rBV A/B-02
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Botulism Vaccine
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 Placebo (Placebo Comparator)
  Interventions: Biological: Placebo (USP sterile saline for injection)
- 2 rBV A/B Vaccine (Active Comparator)
  Interventions: Biological: rBV A/B-40 vaccine
- 3 Placebo (Placebo Comparator)
  Interventions: Biological: Placebo (USP sterile saline for injection)
- 4 rBV A/B Vaccine (Active Comparator)
  Interventions: Biological: rBV A/B-40 vaccine

INTERVENTIONS:
Biological: Placebo (USP sterile saline for injection) — 0.5 mL dose of placebo given by intramuscular injection at Days 0, 28, and 182
  Other Names: placebo
  Arms: 1 Placebo
Biological: rBV A/B-40 vaccine — 0.5 mL dose of rBV A/B-40 vaccine given by intramuscular injection at Days 0, 28 and 182
  Arms: 2 rBV A/B Vaccine
Biological: Placebo (USP sterile saline for injection) — 0.5 mL dose of placebo given by intramuscular injection at Days 0, 56 and 182
  Other Names: placebo
  Arms: 3 Placebo
Biological: rBV A/B-40 vaccine — 0.5 mL dose of rBV A/B-40 vaccine given by intramuscular injection at Days 0, 56 and 182
  Other Names: rBV A/B vaccine
  Arms: 4 rBV A/B Vaccine

SUMMARY:
This Phase 2 study is a double blind, placebo-controlled, randomized, multicenter investigation of rBV A/B-40 vaccine or placebo in healthy adults, using two different three-dose dosing schedules.

DETAILED DESCRIPTION:
The study includes 18 months (547 days) of follow-up after the first vaccination for all randomized volunteers who receive at least one vaccination. Analysis of cumulative data collected through Day 547 ± 14 days will be reported in the final clinical study report.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer has signed the informed consent form.
2. The volunteer is 18 to 55 years of age.
3. The volunteer agrees not to donate blood or blood product for therapeutic or research purposes.
4. The volunteer is willing to comply with the requirements of the protocol.
5. The volunteer has no clinically significant abnormalities on electrocardiogram.
6. Female volunteers of childbearing potential must not be pregnant or lactating and agree to use two types of an acceptable form of FDA-approved contraception through Day 365 ± 7 days.
7. The volunteer is in good health.
8. The volunteer has clinical laboratory test results within the ranges listed in the protocol.

Exclusion Criteria:

1. The volunteer has a history of botulism or prior receipt of any botulinum vaccine, toxoid or antitoxin.
2. The volunteer has previously been treated or expects to be treated with any therapeutic products containing BoNTs such as Botox®, Myobloc®/Neurobloc™ and Botox® Cosmetic.
3. The volunteer has a history of hypersensitivity or significant adverse reaction to other vaccines, aluminum compounds or yeast.
4. The volunteer has donated one or more units of blood or undergone plasmapheresis within the past 28 days.
5. The volunteer received any blood product or immunoglobulin in the previous 6 months.
6. The volunteer received any investigational vaccine in the previous 6 months.
7. The volunteer received any licensed nonliving vaccine within 14 days before or after a scheduled vaccination.
8. The volunteer received any licensed live vaccine within 60 days before or after a scheduled vaccination.
9. The volunteer received any investigational drug therapy within 30 days before the first vaccination or before the last scheduled visit.
10. The volunteer received therapy with immunosuppressive agents, including use of moderate to high-dose oral inhaled or systemic corticosteroids (prednisone-equivalent dose of ≥ 20 mg/day).
11. The volunteer had neurological conditions associated with spasticity or abnormal muscle contraction, demyelination, other abnormalities of smooth or skeletal muscle function, migraine headache, or hyperhidrosis.
12. The volunteer had systemic or recurrent disease or condition that would place the volunteer at an unacceptable risk of injury or requires frequent or continuous medical intervention for treatment, has required hospitalization, or is likely to require surgical intervention during the course of the study.
13. The volunteer has a history of immunodeficiency or autoimmune disease.
14. The volunteer has a systemic medical condition that is ongoing or has required hospitalization or administration of antimicrobial agents within 6 months before screening.
15. The volunteer has a history of arthritis on more than one occasion not related to trauma or any episode of non-trauma-related arthritis within the previous 6 months.
16. The volunteer has an acute self-limited illness that has not resolved by the time of first vaccination including oral temperature greater than 99.5 °F.
17. The volunteer has a history of abuse of alcohol or drugs within the 12 months before study screening.
18. The volunteer has occupational or other responsibilities that would prevent completion of participation in the study.
19. The volunteer has a body mass index ≥ 35 kg/m2.
20. The volunteer has a confirmed positive result on a urine drug screen that tests for common substances of abuse such as amphetamines, barbiturates, benzodiazepines, cocaine, opiates and cannabinoids.
21. The volunteer was seropositive on screening tests for human immunodeficiency virus, hepatitis C virus or hepatitis B surface antigen.
22. The volunteer is currently on active duty in the U.S. military.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary safety objective is to assess rBV A/B-40 vaccine or placebo given to volunteers with an observation period of 30 weeks (Day 210 ± 7 days). The primary immunogenicity objective is to evaluate neutralizing antibody rate. | 30 weeks (Day 210 ± 7 days)

SECONDARY OUTCOMES:
The secondary safety objective is to assess rBV A/B-40 vaccine or placebo given to volunteers with an observation period of 18 months (Day 547 ± 14 days). The secondary immunogenicity objectives include evaluating antibody kinetics. | 18 months (Day 547 ± 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: William Swiderski, Study Director — DynPort Vaccine Company LLC; George A. Saviolakis, M.D., Study Director — DynPort Vaccine Company LLC
Locations (6):
- United States (6):
  - Miami Research Associates, Miami, Florida
  - University Clinical Research, Inc, Pembroke Pines, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Wake Research Associates, Raleigh, North Carolina
  - Clinical Research Associates of Tidewater, Norfolk, Virginia